CLINICAL TRIAL: NCT01333410
Title: Comparison the Efficacy and Safety of 0.1% Tacrolimus Ointment With 0.1% Mometasone Furoate Cream in the Treatment of Adult Vitiligo: A Single Blinded Pilot Study
Brief Title: Comparison of Efficacy and Safety of 0.1% Tacrolimus and 0.1% Mometasone Furoate for Adult Vitiligo
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, chanisada tuchinda, Assistant Professor, Mahidol University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: MahidolU
Record Dates: First submitted 2011-04-08; First posted 2011-04-12 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-10

CONDITIONS: Vitiligo
Keywords: vitiligo; tacrolimus; mometasone furoate
MeSH Terms: conditions — Vitiligo | interventions — Tacrolimus; Mometasone Furoate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 0.1% tacrolimus ointment (Active Comparator)
  Interventions: Drug: tacrolimus ointment
- 0.1% mometasone furoate cream (Active Comparator)
  Interventions: Drug: Mometasone furoate

INTERVENTIONS:
Drug: tacrolimus ointment — 2 applications per days for 6 months
  Other Names: protopic
  Arms: 0.1% tacrolimus ointment
Drug: Mometasone furoate — 2 applications per day for 6 months
  Other Names: elomet
  Arms: 0.1% mometasone furoate cream

SUMMARY:
Vitiligo has remained a difficult disease to treat. Previous available therapies are often ineffective. It usually takes several months or years for complete repigmentation and some areas of the body get at best only partial repigmentation. The desire of the patient to undergo therapy varies from patient to patient and needs to be assessed individually. Several factors should be considered when planning the treatment strategies including type of vitiligo, site and degree of involvement, skin color, psychological effect, patient compliance, ease to assess to therapy, cost of treatment and social association of the disease.

Topical corticosteroids are still be the standard treatment of localized vitiligo. However, the adverse effects such as skin atrophy, striae, pigmentary change and hypothalamic-pituitary adrenal axis suppression can occur if we use inappropriate strength of topical steroids for a long period of time.

Tacrolimus (FK-506) is a new immunosuppressive agent that acts by inhibiting T-cell activation and cytokine release. It offers a safe and efficacious alternative for many skin conditions. It minimizes the need for topical glucocorticoids and does not cause skin atrophy. Tacrolimus was first reported for treatment of vitiligo in 2002. The underlying mechanism was shown in an in vitro study that topical tacrolimus promoted proliferation of melanocytes and melanoblasts.

This study purpose is to evaluate the efficacy and safety of 0.1% topical tacrolimus ointment comparing to 0.1% mometasone furoate cream in the treatment of adult vitiligo.

DETAILED DESCRIPTION:
At first visit, patients will be randomized to receive 0.1% tacrolimus ointment for apply to vitiligo lesion on one side of the body. The lesion on the other side of the body will be treated with 0.1% mometasone furoate cream. Patients are instructed to apply 0.1% tacrolimus ointment and 0.1% mometasone furoate cream twice a day for 6 months

Patients will be follow up at 2, 4 and 6 months for clinical improvement, side effects and photographs

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be above 18 years old
2. Patients must have symmetrical vitiligo lesion on both sides of the body. Total vitiligo area is not exceeded 5% of the body surface area
3. Discontinue any previous systemic medication or phototherapy for at least 3 months and discontinue any topical medication for at least 1 month before starting the study

Exclusion Criteria:

1. Patient who have the lesion on acral area (hands or feet)
2. Pregnancy or lactation patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-06; Primary Completion 2013-06 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
percent of repigmentation | 6 months
  Percent of patients who get repigmentation of the lesion after 0.1% tacrolimus ointment VS 0.1% mometasone furoate cream Percent of repigmentation is defined as following
  * No improvement (0 % repigmentation)
  * Improved by 1-25% repigmentation
  * Improved by 26-50% repigmentation
  * Improved by 51-75% repigmentation
  * Improved by 76-100% repigmentation

SECONDARY OUTCOMES:
side effect | 6 months
  Possible side effect from topical 0.1% tacrolimus ointment and 0.1% mometasone furoate cream

CONTACTS AND LOCATIONS:
Overall Officials: Chanisada Wongpraparut, M.D., Principal Investigator — Siriraj Hospital
Locations (1):
- Department of Dermatology, Faculty of Medicine Siriraj Hospital, Bangkok, Thailand